CLINICAL TRIAL: NCT00448279
Title: A Randomized, Open-label Study to Compare Progression-free Survival in Patients With HER2 Positive Metastatic Breast Cancer Who Continue or Discontinue Herceptin in Combination With 2nd Line Chemotherapy, Having Progressed on 1st Line Chemotherapy in Combination With Herceptin
Brief Title: THOR Study: A Study of Continued Herceptin (Trastuzumab) in Combination With Second Line Chemotherapy in Patients With HER2 Positive Metastatic Breast Cancer.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML18742
Record Dates: First submitted 2007-03-15; First posted 2007-03-16 (Estimated); Results first posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Drug Therapy

ARMS (2):
- Chemotherapy Alone (Active Comparator): Chemotherapy, schedule and dose at the investigator's discretion.
  Interventions: Drug: Chemotherapy
- Chemotherapy, Trastuzumab (Experimental): Trastuzumab, at the investigator's discretion, either 2 milligrams per kilogram (mg/kg) intravenous (i.v.) every 7 days or 6 mg/kg i.v. every 3 weeks. Chemotherapy, schedule and dose at the investigator's discretion.
  Interventions: Drug: trastuzumab; Drug: Chemotherapy

INTERVENTIONS:
Drug: trastuzumab — 2mg/kg i.v. weekly, or 6mg/kg i.v. every 3 weeks
  Other Names: Herceptin
  Arms: Chemotherapy, Trastuzumab
Drug: Chemotherapy — Schedule and dose at the investigator's discretion

SUMMARY:
This 2 arm study will compare the efficacy and safety of continuation or discontinuation of Herceptin treatment in combination with 2nd line chemotherapy, in patients with HER2 positive metastatic breast cancer whose condition has progressed on 1st line chemotherapy plus Herceptin. Patients will be randomized either to continue or discontinue Herceptin treatment (2mg/kg iv infusion weekly, or 6mg/kg iv infusion every 3 weeks) while receiving 2nd line chemotherapy of the investigator's choice. The anticipated time on study treatment is until disease progression, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* female patients, >=18 years of age;
* metastatic breast cancer;
* HER2 overexpression (IHC 3+ and/or FISH positive);
* disease progression during or after previous 1st line chemotherapy plus Herceptin;
* scheduled to receive 2nd line chemotherapy.

Exclusion Criteria:

* incompatibility with previous Herceptin therapy;
* pregnancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (34):
- Italy (34):
  - Avellino
  - Brescia
  - Candiolo
  - Carrara
  - Cona (Ferrara)
  - Cosenza
  - Crotone - Kr
  - Fano
  - Florence
  - Frattaminore
  - Genova
  - Lecce
  - Livorno
  - Mantova
  - Meldola
  - Napoli
  - Nocera Inferiore
  - Padua
  - Palermo
  - Pavia
  - Perugia
  - Pordenone
  - Potenza
  - Ragusa
  - Reggio Calabria
  - Rionero in Vulture
  - Roma
  - Salerno
  - San Giovanni Rotondo
  - Sassari
  - Sora
  - Taormina
  - Torino
  - Udine

RESULTS

PARTICIPANT FLOW:
Groups:
- Chemotherapy Alone: Participants received chemotherapy until disease progression, unacceptable toxicity, or death; the schedule and dose at the investigator's discretion and per local prescribing guidelines and standard center practice. Allowed chemotherapy regimens included paclitaxel, gemcitabine, platinum compounds, docetaxel, capecitabine, or vinorelbine.
- Chemotherapy Plus (+) Trastuzumab: Participants received trastuzumab at either 2 milligrams per kilogram (mg/kg), intravenously (IV), every 7 days, or 6 mg/kg, IV, every 3 weeks, per the investigator's discretion. Participants also received chemotherapy; the schedule and dose at the investigator's discretion and per local prescribing guidelines and standard center practice. Allowed chemotherapy regimens included paclitaxel, gemcitabine, platinum compounds, docetaxel, capecitabine, or vinorelbine. Study treatment was administered until disease progression, unacceptable toxicity, or death.
Period: Overall Study
Arm/Group | Chemotherapy Alone | Chemotherapy Plus (+) Trastuzumab
Started | 29 | 29
Completed | 0 | 0
Not Completed | 29 | 29
Not completed — Lost to Follow-up | 2 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Disease progression | 16 | 18
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Other | 6 | 4
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: all randomized participants.
Groups:
- Chemotherapy + Trastuzumab: Participants received trastuzumab at either 2 mg/kg, IV, every 7 days, or 6 mg/kg, IV, every 3 weeks, per the investigator's discretion. Participants also received chemotherapy; the schedule and dose at the investigator's discretion and per local prescribing guidelines and standard center practice. Allowed chemotherapy regimens included paclitaxel, gemcitabine, platinum compounds, docetaxel, capecitabine, or vinorelbine. Study treatment was administered until disease progression, unacceptable toxicity, or death.
- Total: Total of all reporting groups
Arm/Group | Chemotherapy Alone | Chemotherapy + Trastuzumab | Total
Number analyzed (Participants) | 29 | 29 | 58
Age, Continuous [Median (Full Range); unit: years] | 59 [38 to 81] | 57 [39 to 82] | 58 [38 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) - Percentage of Participants With an Event
Description: PFS was defined as the time from randomization to the date of documented disease progression according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, or the date of occurrence of a second primary cancer, or date of death from any cause, whichever comes first. Participants were censored at the last tumour evaluation.
Time Frame: Baseline (BL) and every 8 weeks thereafter
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy Alone | Chemotherapy + Trastuzumab
Number analyzed (Participants) | 29 | 29
percentage of participants | 58.6 | 58.6

2. Primary Outcome: Progression-Free Survival - Time to Event
Description: The median time from randomization to PFS event. Participants were censored at the last tumour evaluation.
Time Frame: BL and every 8 weeks thereafter
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy Alone | Chemotherapy + Trastuzumab
Number analyzed (Participants) | 29 | 29
months | 9.7 [5.5 to 18.9] | 9.4 [6.7 to 12.0]

3. Secondary Outcome: Overall Survival (OS) - Percentage of Participants With an Event
Description: OS was defined as the time from randomization to the date of death from any cause. Participants were censored at the last contact date at which the participant was known to be alive.
Time Frame: BL and every 8 weeks thereafter
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy Alone | Chemotherapy + Trastuzumab
Number analyzed (Participants) | 29 | 29
percentage of participants | 55.2 | 34.5

4. Secondary Outcome: Overall Survival - Time to Event
Description: The median time from randomization to OS event. Participants were censored at the last contact date at which the participant was known to be alive.
Time Frame: BL and every 8 weeks thereafter
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy Alone | Chemotherapy + Trastuzumab
Number analyzed (Participants) | 29 | 29
months | 19.1 [17.0 to 32.7] | 26.7 [14.0 to NA] — Upper limit of the 95 percent (%) confidence interval (CI) could not be determined as follow-up was too short to observe enough survival events for complete data estimation.

5. Secondary Outcome: Percentage of Participants by Best Overall Response (BOR)
Description: BOR was defined as the best objective response observed during the treatment period according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Complete response (CR): disappearance of all target lesions (TLs), with any pathological lymph nodes (whether target or non-target) having a reduction in short axis to less than 10 millimeters (mm). Partial response (PR): at least a 30 percent (%) decrease in the sum of diameters of TLs, taking as reference the BL sum diameters. Progressive disease (PD): at least a 20% increase in the sum of diameters of TLs, taking as a reference the smallest sum on study (this included the BL sum if that is the smallest on study). In addition to the relative increase in 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. Stable disease (SD) was defined as neither sufficient shrinkages to qualify for PR, nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: BL and every 8 weeks thereafter
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Chemotherapy Alone | Chemotherapy + Trastuzumab
Number analyzed (Participants) | 29 | 29
percentage of participants
  CR | 0 | 10.3
  PR | 27.6 | 20.7
  SD | 24.1 | 24.1
  PD | 17.2 | 13.8
  Not Evaluated | 31.0 | 31.0

6. Secondary Outcome: Percentage of Participants With a Best Overall Response of CR or PR
Description: BOR was defined as the best objective response observed during the treatment period according to RECIST version 1.1. CR: disappearance of all TLs, with any pathological lymph nodes (whether target or non-target) having a reduction in short axis to less than 10 mm. PR: at least a 30% decrease in the sum of diameters of TLs, taking as reference the BL sum diameters. PD: at least a 20% increase in the sum of diameters of TLs, taking as a reference the smallest sum on study (this included the BL sum if that is the smallest on study). In addition to the relative increase in 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. SD: neither sufficient shrinkages to qualify for PR, nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: BL and every 8 weeks thereafter
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy Alone | Chemotherapy + Trastuzumab
Number analyzed (Participants) | 29 | 29
percentage of participants | 27.6 [12.7 to 47.2] | 31.0 [15.3 to 50.8]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded throughout the study. Drug-related serious AEs (SAEs) were collected, regardless of the time elapsed from last study treatment administration, even if the study had been closed.
Description: All randomized participants who received at least 1 dose of study treatment were included in the safety evaluation.
Arm/Group | Chemotherapy Alone | Chemotherapy + Trastuzumab
Serious Adverse Events (participants affected / at risk) | 4/26 | 1/28
Other Adverse Events (participants affected / at risk) | 26/26 | 26/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy Alone (N=26) | Chemotherapy + Trastuzumab (N=28)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
General Malaise (General disorders) | 1 | 0
Gastric volvulus (Gastrointestinal disorders) | 0 | 1
Acute renal failure (Renal and urinary disorders) | 1 | 0
Hospitalisation for intrapleuric chemotherapy and thoracentesis (General disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chemotherapy Alone (N=26) | Chemotherapy + Trastuzumab (N=28)
Leukopenia (Blood and lymphatic system disorders) | 13 | 7
Neutropenia (Blood and lymphatic system disorders) | 16 | 9
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 8 | 1
Mucositis (Gastrointestinal disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 5 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 3
Depression (Psychiatric disorders) | 0 | 1
Liver-GOT,GPT (Hepatobiliary disorders) | 1 | 1
Other - unspecified (General disorders) | 8 | 9
Neuro device (Nervous system disorders) | 0 | 3
Anxiety (Psychiatric disorders) | 0 | 2
Pain (General disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 5
Dysgeusia (Nervous system disorders) | 2 | 0
Cutanea SMP (Skin and subcutaneous tissue disorders) | 1 | 3
Vertigo syndrome (Nervous system disorders) | 1 | 0
Scapular pain (General disorders) | 1 | 1
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Dorsal spine pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Fever (General disorders) | 5 | 3
Vomiting (Gastrointestinal disorders) | 5 | 1
Liver-ALP (Hepatobiliary disorders) | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Asthenia (General disorders) | 7 | 1
Pain - Spine (Musculoskeletal and connective tissue disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Decline in mood (Psychiatric disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Allergy (Immune system disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 2
Heartburn (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 0
Plantar foot pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Exertional dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hand fissures (General disorders) | 1 | 0
Paresthesia - hand (Nervous system disorders) | 1 | 0
Gingival (Gastrointestinal disorders) | 1 | 0
Pelvic pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Memory deficit (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abdominal cramps (Gastrointestinal disorders) | 1 | 0
Epigastric pain (Gastrointestinal disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Sore throat (Gastrointestinal disorders) | 1 | 0
Edema (General disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Urinary infection (Infections and infestations) | 0 | 1
Right upper limb pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cranial pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Paraesthesia hand and feet (Nervous system disorders) | 0 | 1
Achy hands and feet (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Hypercholesterolemia (Investigations) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Bilateral mandibular pain (Gastrointestinal disorders) | 1 | 0
Erythema hand and foot (Skin and subcutaneous tissue disorders) | 1 | 0
Liver-bilirubin (Hepatobiliary disorders) | 0 | 1
Diabetes (Metabolism and nutrition disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.